CLINICAL TRIAL: NCT01806337
Title: Prospective Phase II Study for Treatment Peripheral T-cell Lymphoma, CHOP-14 Plus PEG-Filgrastim Followed by Alemtuzumab Consolidation
Brief Title: CHO(E)P-14 Followed by Alemtuzumab Consolidation in Peripheral T Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Lorenz, Trümper, MD, MD, University of Göttingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL-2003-1; German High Grade Lymphoma SG (Other: DSHNHL)
Record Dates: First submitted 2013-02-25; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Peripheral T-Cell Lymphoma
Keywords: peripheral T cell lymphoma; alemtuzumab; consolidation
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab, antibody (Experimental): alemtuzumab - anti CD 52 antibody administered as consolidation, total dose 133 mg
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Consolidation after CHOP induction
  Other Names: MabCampath

SUMMARY:
Prospective Phase II Study for Treatment Peripheral T-cell Lymphoma, CHOP-14 Plus PEG-Filgrastim Followed by Alemtuzumab Consolidation

DETAILED DESCRIPTION:
Peripheral T cell lymphoma patients of all subtypes according to WHO are treated with an induction of 6 cycles of CHOP-etoposide-14 (if below 60 years of age) oder CHOP-14. If at least a PR is reached, consolidation with alemtuzumab, total dose 133 mg, is given i.v.

ELIGIBILITY:
Inclusion Criteria:

* all risk groups in international prognostic index
* diagnosis of aggressive T-cell-lymphoma, confirmed by an excisional biopsy of a lymph node or by sufficiently extensive biopsy of an extranodal involvment, if there is no lymph node involvment.
* these lymphomas comprise: peripheral T-cell lymphoma PTCL-NOS Lennert´s lymphoma T-zone lymphoma angioimmunoblastic T-cell-lymphoma
* Performance status: ECOG (Eastern Cooperative Oncology Group Score) 0-3(Karnofsky index 40-100%)
* written consent of the patient
* Declaration of center participation

Exclusion Criteria:

* Already initiated lymphoma therapy(exept for the prephase treatment specified for this study)
* Serious accompanying disorder or impaired organ function
* bone marrow involvement>25%
* Known hypersensitivity to medications to be used
* Know HIV-positivity
* Active hepatitis infection, active CMV infection, prior florid tuberculosis
* floride systemic infections
* suspicion that patient compliance will be poor
* Simultaneous participation in any the study protocol
* prior chemo-or radiotherapy for malignancy
* other concomitant malignant disease
* Pregnancy or lactation period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-07; Primary Completion 2006-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of alemtuzumab consolidation after CHO(E)P 14 induction chemotherapy | average of 24 weeks (treatment duration)
  A descriptive approach for the primary endpoint was chosen: Adherence to schedule of alemtuzumab consolidation (number of cycles, dosing, time) - comparison of planned vs given in pts receiving alemtuzumab

SECONDARY OUTCOMES:
rate of complete remissions | at week 24 after initiation
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Truemper, Principal Investigator — German High Grade Non Hodgkin´s Lymphoma Study Group